CLINICAL TRIAL: NCT00895076
Title: A Randomized, Open-Label, Single Dose, Two-Way Crossover Study to Evaluate the Pharmacokinetics and Safety of a Dexamethasone Iontophoretic Transdermal Patch Compared to Dexamethasone Injection in Healthy Adult Volunteers
Brief Title: Study to Compare the Pharmacokinetics of a Dexamethasone Iontophoretic Patch to a Dexamethasone Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Travanti Pharma Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Robert Cooper, M.D. / Principle Investigator, Cetero Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
MeSH Terms: conditions — Tennis Elbow | interventions — Dexamethasone

ARMS (2):
- 1 (Experimental): dexamethasone iontophoretic patch
  Interventions: Drug: dexamethasone
- 2 (Active Comparator): dexamethasone intramuscular injection
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — iontophoretic patch and injection

SUMMARY:
The primary objectives are to evaluate the extent of systemic exposure and dexamethasone bioavailability following a single application of a dexamethasone iontophoretic transdermal patch in healthy volunteers.

The secondary objectives are to evaluate the systemic and topical safety of the dexamethasone iontophoretic transdermal patch and of the dexamethasone intramuscular (IM) injection.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 Years to 45 Years
* Must have a Body Mass Index (BMI) between 18 and 29 kg/m2, inclusive.
* Must, in the investigator's opinion, have no clinically significant disease as determined by medical and psychiatric history, physical examination, vital signs, and/or laboratory evaluations conducted at the screening visit or on clinic admission that would interfere with the evaluation of safety or pharmacokinetics.
* Must have negative screens for Hbs-Ag, HCV-Ab, and HIV-Ab, and no history of a positive result.
* Female subjects may be included if they are surgically sterile or 2 years post menopausal, and they have a negative serum pregnancy test at screening. Female subjects of child bearing potential and peri-menopausal subjects may be included if they have a negative serum pregnancy test at screening and on admission to the clinic on Day -1, and agree to use a medically accepted method of birth control (e.g., barrier method with spermicide, oral contraceptive, or abstinence) and agree to continue use of this method for the duration of the trial.
* Must be non-smokers, defined as not having smoked tobacco, used chewing tobacco, or used nicotine-containing products for smoking cessation in the 6 months prior to screening.
* Must be able to communicate effectively with the study personnel.
* Must agree to remain in the study facility overnight for approximately five consecutive days and nights.

Exclusion Criteria:

* Is a female subject who is pregnant, breastfeeding, or planning a pregnancy during the study.
* Has a clinically significant unstable medical abnormality, chronic disease, significant neurological (including seizure and cognitive disorders), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease, or any other abnormality that could interfere with the PK evaluation of the study drug. Particular attention will be paid to exclude subjects with a risk for the consequences of systemic corticosteroid exposure, such as diabetes or poorly controlled hypertension.
* Has had a clinically significant illness within 30 days of Screening.
* Use of any prescription medication (other than hormonal contraceptives) within 14 days or over-the-counter (OTC) medication (with the exception of ibuprofen and acetaminophen) within 7 days of randomization or intends to use any prescription or OTC medication during the study that may interfere with the evaluation of the study drug.
* Use of any topical creams, lotions or oils on the patch application site within 2 weeks of treatment administration in the first period and throughout the study.
* Use of any steroid, including topical steroid, within 4 weeks of treatment administration in the first period and throughout the study.
* Intake of grapefruit products, and foods, herbal products and over-the-counter or prescription medications that may interact with the CYP450 enzyme system from 7 days prior to treatment administration in the first period until completion of the end-of-study procedures.
* Has ingested alcohol within 24 hours before admission (Day -1) and throughout the study.
* Has a history of significant allergy or hypersensitivity to the study drugs or to any component of iontophoretic transdermal patch used in this study, including allergy or sensitivity to bandage adhesives or to sodium bisulfate.
* Has any of the following exclusionary clinical laboratory results:

  1. Hemoglobin less than 12.0 g/dL
  2. Serum creatinine greater than 2.0 mg/dL
  3. Abnormal liver function tests (serum glutamic oxaloacetic transaminase [SGOT], also called aspartate transaminase [AST]; or serum glutamic pyruvic transaminase [SGPT], also called alanine transaminase [ALT] more than twice the upper limit of normal)
  4. Elevated serum bilirubin more than 2 times the upper limit of normal
* Any blood donation or significant blood loss within 90 days of treatment administration in the first period.
* Any plasma donation within 7 days of randomization.
* Has any sensory dysfunction, any skin irritation, sensitivity or disease, or a tattoo that may in the opinion of the investigator interfere with assessment of topical effects at the site of patch application.
* Has history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of study enrollment.
* Has or develops a positive urine drug screen, including ethanol, cocaine, tetrahydrocannabinol, barbiturates, amphetamines, benzodiazepines, and opiates.
* Use of any other investigational drug within 30 days or five half-lives (whichever is longer) before treatment administration in the first period, or plans to use an investigational drug (other than the study drugs) during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
The primary objectives are to evaluate the extent of systemic exposure and dexamethasone bioavailability following a single application of a dexamethasone iontophoretic transdermal patch in healthy volunteers. | 0-33 hours
Pharmacokinetics and safety of dexamethasone iontophoretic patch | 0-33 hours

SECONDARY OUTCOMES:
The secondary objectives are to evaluate the systemic and topical safety of the dexamethasone iontophoretic transdermal patch and of the dexamethasone IM injection. | 0-33 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Research, Fargo, North Dakota, United States